CLINICAL TRIAL: NCT02788058
Title: A Phase II Trial of Hypofractionated Radiotherapy for Limited Metastatic NSCLC Harboring Sensitizing EGFR Mutations After First Line TKI Therapy
Brief Title: A Study of Hypofractionated Radiotherapy for Limited Metastatic NSCLC Harboring Sensitizing EGFR Mutations After First Line TKI Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZCH-2016-08
Record Dates: First submitted 2016-04-22; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Lung Adenocarcinoma; EGFR Positive Non-small Cell Lung Cancer
Keywords: Hypofractionated Radiotherapy; EGFR Positive; Lung Adenocarcinoma; Limited Metastases
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGFR-TKI (Experimental): Patients take EGFR-TKI alone till tumor progression
  Interventions: Drug: EGFR-TKI
- EGFR-TKI+hypofractionated radiotherapy (Active Comparator): After 3 mos TKI, patients with limited metastatic take EGFR-TKI concurrent with hypofractionated radiotherapy till tumor progression.
  Interventions: Drug: EGFR-TKI; Radiation: Thoracic Hypofractionated Radiotherapy

INTERVENTIONS:
Drug: EGFR-TKI — Gefitinib 250mg po qd or Erlotinib 150mg po qd or Icotinib 125mg po tid
  Other Names: Gefitinib/Erlotinib/Icotinib
Radiation: Thoracic Hypofractionated Radiotherapy — 40-45 Gy/5-15f
  Arms: EGFR-TKI+hypofractionated radiotherapy

SUMMARY:
To evaluate the efficacy and toxicity of patients treated with hypofractionated radiotherapy for limited metastatic NSCLC harboring sensitizing EGFR mutations after first line TKI therapy. An exploratory biomarker analysis in blood and tumor samples is also planned.

DETAILED DESCRIPTION:
Rational:

After inductive TKI therapy in NSCLC with sensitizing EGFR mutations, the residual lesion might be the source of subsequent disease progression, defined as acquired resistance to TKI. Two reasons can be used to explain the formation of the residual lesion：1）there is a subgroup of cancer cells that are not sensitive to TKI therapy because of tumor heterogeneity, like de novo T790M mutation; 2)some cancer cells can keep static state during the beginning treatment, and then develops acquired resistance to TKI therapy under the long-term drug pressure and continue to re-proliferation. From this point of view, elimination of residual lesion provides the chance to reduce or slow the possibility of developing resistance to TKI.

Objective:

To evaluate the efficacy and toxicity of patients treated with hypofractionated radiotherapy for limited metastatic NSCLC harboring sensitizing EGFR mutations after first line TKI therapy. An exploratory biomarker analysis in blood and tumor samples is also planned.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic lung adenocarcinoma harboring sensitizing EGFR mutations (L858R, exon 19 deletion), and became oligometastatic disease after 3 months TKI, evaluated by PET/CT scan, brain MRI, and abdomen ultrasound (≤6 discrete lesions of disease, exclusive of the brain metastases, ≤3 lesions in the liver, ≤3 lesions in the lung);
* All sites of disease must be amenable to definitive RT;
* An intrathoracic lymph nodal station is considered 1 discrete lesion, according to IASLC lymph nodal station map;
* Age 18 years or older;
* ECOG Performance Status 0-2;
* Adequate bone marrow, liver and renal function, as specified below: Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L; Hemoglobin ≥ 8 g/dL; Platelets ≥ 100 x 109/L; Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) ; AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present; Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal;
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting treatment;
* Men and women of childbearing age must be willing to use effective contraception while on treatment and for at least 3 months thereafter;
* Patients and their family signed the informed consents;

Exclusion Criteria:

* Received chemotherapy before TKI therapy;
* Brain parenchyma or leptomeningeal disease;
* Any site of disease that is not amenable to definitive RT;
* Concurrent malignancies other than non-melanoma skin cancer that require active ongoing treatment;
* Any medical co-morbidities that would preclude radiation therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-05; Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 years

SECONDARY OUTCOMES:
Frequency of T790M mutation before treatment detected by ctDNA | 1 months
Abundance of T790M mutation before treatment detected by ctDNA | 1 months
Frequency of T790M mutation after radiotherapy detected by ctDNA | 3 months
Abundance of T790M mutation after radiotherapy detected by ctDNA | 3 months
Frequency of T790M mutation after 1 year detected by ctDNA | 1 year
Abundance of T790M mutation after 1 year detected by ctDNA | 1 year
Rate of CTCAE grade 2 or higher radiation pneumonitis | 1 years
  We will assess the rate of symptomatic radiation pneumonitis in patients who received the radiation therapy.
To assess the short-term quality of life (QOL) | 4 months
  FACT-E score at the 4 months after docetaxel consolidation therapy